CLINICAL TRIAL: NCT02642770
Title: 3D & Speckle Tracking Together as a Sensitive Marker for Early Outcome in Patients With Left Ventricular Dysfunction Undergoing Cardiac Surgery
Brief Title: 3D & Speckle Tracking Together as a Marker for Early Outcome in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr Alok Kumar, Fellow, Cardiac Anaesthesia, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: NK/2440/DM/2266
Record Dates: First submitted 2015-12-26; First posted 2015-12-30 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Left Ventricular Systolic Dysfunction
Keywords: Transesophageal echocardiography, Speckle tracking strain
MeSH Terms: conditions — Ventricular Dysfunction, Left | interventions — Echocardiography, Transesophageal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Transesophageal echocardiography — 2D LV Speckle tracking strain and 3D LVEF measurements

SUMMARY:
Patients presenting with Left Ventricle (LV) dysfunction undergoing cardiac surgery are at increased risk of perioperative morbidity and mortality. LV dysfunction has been reported as an independent predictor of operative mortality in patients undergoing Cardiac surgery. It also often leads to low cardiac output states with many of these patients requiring inotropic or mechanical support and vasopressors for hours to days after surgery. Speckle tracking when combined with three dimensional (3D) imaging techniques might prove to be a more sensitive marker for ventricular dysfunction. The present study investigates early outcomes in a consecutive series of patients with LV dysfunction undergoing cardiac surgery

DETAILED DESCRIPTION:
All patients inside operating room, a wide bore i/v access and radial artery will be cannulated under local anesthesia. Standard opioid- propofol- relaxant based induction will be followed. After endotracheal intubation, an adult 2D Trans Eesophageal Echocardiography (TEE) probe (6VT-D probe of the GE vivid E9 echocardiography system (GE Medical Systems, Hortein, Norway) will be inserted. A 7 Fr triple lumen catheter and 8.5 Fr introducer sheath will be placed in the right internal jugular vein under ultrasound guidance. A 7 Fr Pulmonary Artery Catheter (PAC) (Swan Ganz catheter, Edwards Life Sciences) will be floated as per standard practice. Attempts to wedge will be discontinued if the catheter does not wedge beyond 8 cm into the main pulmonary artery.

Surgery will be performed through a midline sternotomy on cardiopulmonary bypass with bicaval cannulation and with intermittent antegrade warm blood cardioplegia. All surgical procedures were performed by experienced surgeons using standardized techniques.

Cardiopulmonary bypass (CPB) and anaesthesia management will be performed according to our standard operating procedures. Moderate hypothermic (28-32*C) CPB will be established with a non-pulsatile flow of 2,5 l/min/m2 and an arterial pressure > 60 mmHg without additional filtration. CPB will be primed with balanced electrolyte solution. Coagulation will be offset by 400 IU/kg heparin aiming at an Activated Clotting Time (ACT) > 480 seconds. Additionally, all patients will receive tranexamic acid 100mg/kg. Cardioplegic arrest will be induced and maintained by intermittent administration of ante grade potassium enriched solution.

Perioperative goal-oriented haemodynamic support (i.e. heart rate 80-100 beats/min, mean arterial pressure 65-85 mmHg, central venous pressure (CVP) 8-12 mmHg at positive end-expiratory pressure 5 cms of water, pulmonary artery occlusion pressure 12-15 mmHg, cardiac index >2.5 l /min/m2 2, stroke volume index >30 ml/m, mixed venous oxygen saturation >65) will be established according to institutional standards. Intraoperatively, patients will be monitored with transoesophageal echocardiography (6VT-D probe of the GE vivid E9 echocardiography system (GE Medical Systems, Hortein, Norway)) and a pulmonary artery catheter with or without continuous mixed venous oximetry measurement. In case of difficult CPB separation despite hemodynamic optimization, an intraaortic balloon pump (IABP) will be placed according to the team's assessment.

After chest closure, the patient will be transferred intubated and mechanically ventilated in the ICU. Patients will be kept sedated with morphine administration (20-40 mcg/kg/min) until cardiopulmonary stability is achieved, chest tube drainage is negligible (<100 ml/h), and the patient is judged to be extubated. If mechanical ventilation is required > 12 hours, sedation will be switched to midazolam (10-20 mcg/kg/min) combined with morphine (20-40 mcg/kg/min), and weaning from mechanical ventilation will be performed according to the standard operating procedures at our hospital. Hemodynamic optimization will be continuously accomplished according to the haemodynamic goals as mentioned above.

The decision for renal replacement therapy (RRT) will be taken in consultation with the department of nephrology and based on the following criteria: a) oliguria < 500 ml/dl and/or anuria < 100 ml/dl, b) metabolic acidosis, c) hyperkaliaemia, and d) uraemia.

Hemodynamic monitoring Once PAC is placed, baseline parameters will be recorded in mmHg. Pressure will be defined as Pulmonary systolic pressure peak (PAPs), mean pressure (PAPm), and Pulmonary Artery Wedge Pressure (PAWP).

These reading will be taken as baseline after placement of PAC. In addition usual vital parameters such as mean blood pressure (MAP), CVP and heart rate (HR), will also be acquired.

Systemic Vascular Resistance (SVR) and Cardiac Index (CI) calculation will be done as per the standard protocol.

Time periods at which parameters will be evaluated After induction of anesthesia hemodynamic and echocardiographic parameters will be taken. After induction, if the patients require ionotropes and/or vasopressors it will be administered to achieve the haemodynamic goal as mentioned above. The parameters will be obtained again after coming out of CPB. Patient will be started on vasopressors- inotropic support as deemed fit by the treating anaesthesiologist to achieve the haemodynamic goal.

End point of study: Either patient dies or discharged from the ICU as per the protocol.

Echocardiographic monitoring All patients in whom TEE probe is placed will undergo an initial comprehensive TEE examination covering all the 28 standard views as per the American Society of Echocardiography (ASE) guidelines. In addition, focused assessment for the study parameters will be done after the completion of comprehensive examination.

Assessment of LV Comprehensive echocardiography will be performed before surgery using 6VT-D probe of the GE vivid E9 echocardiography system (GE Medical Systems, Hortein, Norway), including standard 2D views digitally stored at a high frame rate (>50 frames/s). All measurements will be performed on line on the same machine by anaesthesiologist experienced in TEE blinded to patient's outcome. Left ventricle (LV) volumes in systole and diastole and LV Ejection Fraction (LVEF) will be computed using the Simpson biplane method from 2 chamber (2C) and 4 chamber (4C) apical views. The endocardial borders will be traced for the measurements and the papillary muscles will be excluded, as recommended in the guidelines. A frame rate of >50 will be ensured during the measurements to ensure accurate endocardial border detection. Foreshortening will be avoided by retroflexing the probe.

Speckle-tracking analysis will be performed to assess LV Global Longitudinal strain (GLS). GLS will be computed using 2D-speckle-tracking analysis by automated function imaging (AFI) measured from the three mid esophageal views (long-axis and two- and four-chamber views). For strain processing, the peak of the R-wave on the electrocardiogram will be used as the reference time point for end-diastole and segments with poor-quality tracking will be manually discarded. GLS will only be computed from patients with >14 segments adequately tracked for a 18-segment model. GLS will be calculated by averaging the peak strain values of 18 segments. Three-dimensional LV volumes and EF will be measured from the 3D full-volume data set. Using the on board GE software (GE vivid E9 echocardiography system (GE Medical Systems, Hortein, Norway), the full-volume data of the LV will be organized into orthogonal four-, two-chamber, and short-axis views. Enddiastolic and end-systolic frames will be selected. Mitral annular and apical points will be placed on these images by adjusting the axis. Semi-automated LV endocardial border detection software on the system will outline the endocardial borders in these three planes. The software then uses sequence analysis to track the endocardium in all frames and then automatically calculate a true 3D end diastolic volume (EDV), end systolic volume (ESV), and EF from the moving 3D endocardial shell. The endocardial borders could be adjusted manually if the endocardial border tracking is deemed inadequate, and the sequence analysis will be repeated.

The diastolic function of the LV will be measured by measuring these parameters- the mitral inflow velocity and the tissue Doppler velocity of the lateral mitral annulus. The mitral inflow velocities (E & A) will be measured by placing the cursor for pulsed wave Doppler at the tip of the mitral leaflet coaptation point. The sweep speed will be set at 25mm/s and the scale will be adjusted and the baseline shifted above to obtain optimal waveforms. Tissue Doppler measurements will be taken by placing the cursor of pulsed wave tissue Doppler on the lateral mitral annulus. A frame rate of > 100m/s will be ensured by adjusting the sector width and the measurements made at a sweep aped of 25mm/s.

Post valve replacements, the prosthetic valves will be evaluated as per recommendations for evaluation of prosthetic valves. For all measurements of pulsed and continuous wave doppler the cursor will be placed at an angle < 20' to the flow.

Every attempt will be made to make measurements in sinus rhythm. In case of a non-sinus rhythm, measurements will be taken at the time when the ventricular rate is close to the baseline. If that is not possible, then an average of 5-6 readings will be used for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18yrs) with moderate to severe LV dysfunction (EF< 50%) planned for Coronary artery bypass graft (CABG) and/or valve repair/replacement, presenting to our center for elective or emergent surgery will be included in the study.

Exclusion Criteria:

1. Hypertrophic cardiomyopathy
2. Sepsis
3. Preoperative renal impairment (serum creatinine 2.0 mg/ dL)
4. Off pump CABG
5. Redo surgery.
6. Failed placement despite 3-4 attempts.
7. Congenital heart lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with left ventricular dysfunction (LVEF< 50%) undergoing cardiac surgery under CPB.
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2015-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
incidence of Low Cardiac Output Syndrome | 48 hrs
  Vassopressors Ionotropic Score (VIS) ≥ 15 (> 30 mins) or Requirement of Intra aortic balloon counterpulsation (IABP) in Intensive Care Unit.

SECONDARY OUTCOMES:
Duration of Mechanical Ventilation or Mortality | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: GD Puri, Prof, Study Chair — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- PGIMER, Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ding W, Ji Q, Shi Y, Ma R. Predictors of low cardiac output syndrome after isolated coronary artery bypass grafting. Int Heart J. 2015;56(2):144-9. doi: 10.1536/ihj.14-231. Epub 2015 Feb 23. PMID 25740396